CLINICAL TRIAL: NCT02209909
Title: Effects of Low Dose Aspirin Pre-treatment on Platelet Activation Undergoing Off-pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: OPCAB_ASA_PLT activation
Record Dates: First submitted 2014-07-31; First posted 2014-08-06 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: preoperative aspirin use; platelet activation; off pump coronary artery bypass
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspirin continuation (Experimental): Intervention : Low-dose aspirin (< 100mg/day) is used before OPCAB surgery in the aspirin continuation group.
  Interventions: Drug: aspirin continuation
- aspirin discontinuation (Experimental): Intervention: Low-dose aspirin is stopped more than 4 days before OPCAB surgery in the aspirin discontinuation group.
  Interventions: Drug: aspirin discontinuation

INTERVENTIONS:
Drug: aspirin continuation — Patients are randomized to continue aspirin before OPCAB surgery.
  Other Names: Low-dose aspirin (< 100mg/day)
  Arms: aspirin continuation
Drug: aspirin discontinuation — Patients are randomized to discontinue aspirin more than 4 days before OPCAB surgery.
  Arms: aspirin discontinuation

SUMMARY:
Platelet activation after off pump coronary artery bypass (OPCAB) surgery may affect thrombus formation. The purpose of this study is to assess the effects of preoperative continuation of aspirin on platelet activation after off pump coronary artery bypass surgery.

DETAILED DESCRIPTION:
Patients undergoing OPCAB surgery will be randomized to continue preoperative aspirin or discontinue aspirin before surgery.

Platelet activation can be evaluated by measuring platelet p-selectin using flowcytometry. In this study, we will compare platelet-activated markers and conventional coagulation tests.

ELIGIBILITY:
Inclusion Criteria:

* age : 20-80
* elective OPCAB
* informed consent

Exclusion Criteria:

* coagulation disorder
* emergency operation, re-operation
* co-existing valvular disease
* less than 6 months after cerebral vascular accident
* heparin induced thrombocytopenia
* heparin resistance
* menstrual phase
* preoperative cardiopulmonary bypass, continuous veno-veno hemofiltration, intra-aortic balloon pump application
* less than 12 months after myocardiac infarction
* less than 10 days after unstable angina
* less than 30 days after percutaneous coronary intervention
* less than 6 wks after bare metal stent insertion
* less than 12 months after drug eluting stent insertion

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
change from baseline in platelet p-selectin at 48 hours after operation | after induction of anesthesia(baseline), at the time of end of operation, 24 hour after operation, 48hr after operation
  Primary outcome is expression of platelet p-selectin measured by flowcytometry 48 hours after OPCAB surgery in both groups.

SECONDARY OUTCOMES:
change from baseline in conventional coagulation tests at the time of end of operation, 24 hour after operation, and 48hr after operation | after induction of anesthesia(baseline), at the time of end of operation, 24 hour after operation, 48hr after operation
  prothrombin time (international normalized ratio), activated partial thromboplastin time, fibrinogen

OTHER OUTCOMES:
change from baseline in platelet aggregation at the time of end of operation, 24 hour after operation, and 48hr after operation | after induction of anesthesia(baseline), at the time of end of operation, 24 hour after operation, 48hr after operation
  prediction for stratification of bleeding risk due to antiplatelet agent using multiplate

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea